CLINICAL TRIAL: NCT00108745
Title: A Randomized Phase III Trial of Maintenance Chemotherapy Comparing 12, Monthly Cycles of Single Agent Paclitaxel or CT-2103 Versus No Treatment Until Documented Relapse in Women With Advanced Ovarian, Primary Peritoneal or Fallopian Tube Cancer Who Achieve a Complete Clinical Response to Primary Platinum/Taxane Chemotherapy
Brief Title: Paclitaxel, Polyglutamate Paclitaxel, or Observation in Treating Patients With Stage III or Stage IV Ovarian Epithelial, Peritoneal Cancer, or Fallopian Tube Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0212; NCI-2009-00586 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 07-117; CDR0000422427; GOG-0212; GOG-0212 (Other: NRG Oncology); GOG-0212 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2005-04-18; First posted 2005-04-19 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Ovarian Brenner Tumor; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms | interventions — Watchful Waiting; Observation; Paclitaxel; Taxes; paclitaxel poliglumex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (paclitaxel poliglumex) (Experimental): Patients receive polyglutamate paclitaxel IV over 10-20 minutes on day 1.Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel Poliglumex; Procedure: Quality-of-Life Assessment
- Arm II (paclitaxel) (Active Comparator): Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Procedure: Quality-of-Life Assessment
- Arm III (observation) (Other): Patients receive no further anticancer treatment until evidence of disease progression.
  Interventions: Other: Clinical Observation; Other: Laboratory Biomarker Analysis; Procedure: Quality-of-Life Assessment

INTERVENTIONS:
Other: Clinical Observation — Undergo observation
  Other Names: observation
  Arms: Arm III (observation)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm II (paclitaxel)
Drug: Paclitaxel Poliglumex — Given IV
  Other Names: CT-2103; CT2103; Paclitaxel Polyglutamate; Paclitaxel-Polyglutamate Polymer; PG-TXL; Poly-L-Glutamic acid-Paclitaxel Conjugate; Polyglutamic Acid Paclitaxel; Xyotax
  Arms: Arm I (paclitaxel poliglumex)
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies paclitaxel to see how well it works compared to polyglutamate paclitaxel or observation only in treating patients with stage III or stage IV ovarian epithelial, peritoneal cancer, or fallopian tube cancer. Drugs used in chemotherapy, such as paclitaxel and polyglutamate paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Paclitaxel and polyglutamate paclitaxel may also stop the growth of ovarian epithelial or peritoneal cancer by blocking blood flow to the tumor. Sometimes, after treatment, the tumor may not need additional treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether paclitaxel is more effective than polyglutamate paclitaxel or observation only in treating ovarian epithelial, peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether CT-2103 (polyglutamate paclitaxel) or paclitaxel, administered to women with advanced ovarian, primary peritoneal or fallopian tube cancer who have attained a clinically-defined complete response to primary platinum/taxane-based chemotherapy ("consolidation/maintenance therapy") will reduce the death rate, compared to re-treatment at the time of documented disease progression.

II. To determine if, in this clinical setting, CT-2103 produces a more favorable toxicity profile (with a particular focus on peripheral neuropathy as measured by the Gynecologic Oncology Group [GOG] NTX4) and superior quality-of-life (as measured by the Functional Assessment of Cancer Therapy-Ovarian [FACT-O]), compared to paclitaxel.

SECONDARY OBJECTIVES:

I. To explore the relationship between expression of several of the angiogenic markers and overall survival or progression-free survival in patients randomized to CT-2103, paclitaxel, or no treatment.

II. To assess the association among the various tissue and serum markers of angiogenesis, and compare the ability of different combinations of these markers to predict patient outcome including overall survival and progression-free survival in patients randomized to CT-2103, paclitaxel, or no treatment.

III. To bank deoxyribonucleic acid (DNA) from whole blood for research and evaluate the association between single nucleotide polymorphisms (SNPs) and measures of clinical outcome including overall survival, progression-free survival and adverse events.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive polyglutamate paclitaxel intravenously (IV) over 10-20 minutes on day 1.

ARM II: Patients receive paclitaxel IV over 3 hours on day 1.

ARM III: Patients receive no further anticancer treatment until evidence of disease progression.

In arms I and II, treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of primary peritoneal carcinoma, or stage III or IV epithelial ovarian or fallopian tube carcinoma, with either optimal (=< 1 cm residual disease) or suboptimal residual disease following initial surgery; all patients must have had appropriate surgery for ovarian, primary peritoneal or fallopian tube carcinoma with appropriate tissue available for histologic evaluation to confirm diagnosis and stage
* Patients with the following histologic epithelial cell types are eligible:

  * Serous adenocarcinoma
  * Endometrioid adenocarcinoma
  * Mucinous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial carcinoma
  * Transitional cell carcinoma
  * Malignant Brenner tumor
  * Adenocarcinoma not otherwise specified (NOS)
* Patients must have completed treatment within the past 12 weeks with at least 5 cycles and not more than 8 cycles of a platinum (IV or intraperitoneal [IP]) and paclitaxel or docetaxel-based combination chemotherapy and have no symptoms suggestive of persistent cancer, normal (no evidence of cancer) computed tomography (CT) scan of the abdomen/pelvis and normal cancer antigen 125 (CA-125) following this therapy

  * Patients treated with neo-adjuvant platinum-taxane chemotherapy for a presumptive diagnosis of stage III or IV epithelial ovarian, primary peritoneal or, fallopian tube (by paracentesis, percutaneous biopsy or open biopsy) are eligible provided that they have undergone interval abdominal surgery after at least one but no more than six cycles of standard chemotherapy; such surgery must meet the same criteria as for those undergoing up front surgery, including tissue diagnosis for confirmation of primary tumor site and stage III or IV disease; also, patients must have received at least two cycles after interval abdominal surgery
* Absolute neutrophil count >= 1,500/ul, equivalent to Common Toxicity Criteria (CTCAE version [v]3.0) grade 1
* Platelet count >= 100,000/ul
* Creatinine =< 1.5 times institutional upper limit of normal (ULN), CTCAE v3.0 grade 1
* Bilirubin =< 1.5 times ULN, (CTCAE v3.0 grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) =< 2.5 times ULN (CTCAE v3.0 grade 1)
* Alkaline phosphatase =< 2.5 times ULN (CTCAE v3.0 grade 1)
* Neuropathy (sensory and motor) less than or equal to CTCAE v3.0 grade 1
* Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2
* Patients must have signed an approved informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization
* Patients must complete pre-entry assessments

Exclusion Criteria:

* Patients with a current diagnosis of epithelial ovarian or fallopian tube tumor of low malignant potential (LMP) (Borderline carcinomas) are not eligible; patients with a prior diagnosis of a low malignant potential tumor that was surgically resected and who subsequently develop invasive adenocarcinoma are eligible, provided that they have not received prior chemotherapy for their ovarian LMP tumor
* Germ cell tumors, sex cord-stromal tumors, carcinosarcomas, mixed mullerian tumors or carcinosarcomas, metastatic carcinomas from other sites to the ovary and low malignant potential tumors including so called micropapillary serous carcinomas are not eligible
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than 3 years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received investigational therapies, and/or biological therapies (i.e. Bevacizumab or Erlotinib) for their epithelial ovarian, primary peritoneal or fallopian tube cancers or for any other abdominal or pelvic tumor, are not excluded; however, biologics cannot be continued concurrent with the GOG-012 maintenance treatment (or observation); patients who have received prior chemotherapy for any other abdominal or pelvic tumor (except as noted above) are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than 3 years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded, unless all of the following conditions are met:

  * Stage not greater than I-B
  * Less than 3 mm invasion without vascular or lymphatic invasion
  * No poorly differentiated subtypes, including papillary serous, clear cell, or other Federation of Gynecology and Obstetrics (FIGO) Grade 3 lesions
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy are excluded
* Patients with acute hepatitis, or known chronic hepatitis
* Patients with an active infection that requires antibiotics
* Patients with ongoing gastrointestinal bleeding requiring blood product support
* Patients whose circumstances at the time of entry onto the protocol would not permit completion of study or required follow up
* Patients with unstable angina or those who have had a myocardial infarction within the past six months; patients with evidence of abnormal cardiac conduction (e.g. bundle branch block, heart block) are eligible if their disease has been stable for the past six months
* Patients are excluded who have had prior therapy with CT-2103
* Patients with active bleeding or an unexplained prothrombin time (PT) or partial thromboplastin time (PTT) > institutional upper limit normal (ULN)
* Patients who are pregnant or nursing are excluded; patients who may become pregnant must practice an effective method of birth control

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1157 (Actual)
Dates: Start 2005-03-21 (Actual); Primary Completion 2015-02-03 (Actual); Study Completion 2022-02-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Larry J Copeland, Principal Investigator — NRG Oncology
Locations (315):
- United States (315):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Tennessee Valley Gynecologic Oncology, Huntsville, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Highlands Oncology Group PA - Fayetteville, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Southeast Gynecologic Oncology Associates, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Hospital Medical Center of Queens, Fresh Meadows, New York
  - Queens Hospital Center, Jamaica, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Westchester Medical Center, Valhalla, New York
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Chattanooga Gynecological Oncology, Chattanooga, Tennessee
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - Knoxville Gynecologic Cancer Specialists PC, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Bon Secours Mary Immaculate Hospital, Newport News, Virginia
  - Virginia Oncology Associates - Lake Wright, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Slinger, Slinger, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

REFERENCES:
- [Derived] Copeland LJ, Brady MF, Burger RA, Rodgers WH, Huang HQ, Cella D, O'Malley DM, Street DG, Tewari KS, Bender DP, Morris RT, Lowery WJ, Miller DS, Dewdney SB, Spirtos NM, Lele SB, Guntupalli S, Ueland FR, Glaser GE, Mannel RS, DiSaia PJ. Phase III Randomized Trial of Maintenance Taxanes Versus Surveillance in Women With Advanced Ovarian/Tubal/Peritoneal Cancer: A Gynecologic Oncology Group 0212:NRG Oncology Study. J Clin Oncol. 2022 Dec 10;40(35):4119-4128. doi: 10.1200/JCO.22.00146. Epub 2022 Jun 27. PMID 35759733

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Paclitaxel Poliglumex) | Arm II (Paclitaxel) | Arm III (Observation)
Started | 387 | 384 | 386
Completed | 353 | 349 | 349
Not Completed | 34 | 35 | 37
Not completed — Withdrawal by Subject | 19 | 12 | 12
Not completed — Never Treated | 8 | 10 | 12
Not completed — Ineligible | 7 | 13 | 13

BASELINE CHARACTERISTICS:
Population: All enrolled patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel Poliglumex) | Arm II (Paclitaxel) | Arm III (Observation) | Total
Number analyzed (Participants) | 387 | 384 | 386 | 1157
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.02 (10.89) | 58.80 (10.42) | 59.07 (9.68) | 58.96 (10.34)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 21 | 13 | 11 | 45
  40 - 49 years | 54 | 71 | 57 | 182
  50 - 59 years | 115 | 114 | 138 | 367
  60 - 69 years | 137 | 132 | 126 | 395
  70 - 79 years | 56 | 46 | 49 | 151
  >= 80 years | 4 | 8 | 5 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 387 | 384 | 386 | 1157
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 25 | 16 | 59
  Not Hispanic or Latino | 341 | 338 | 346 | 1025
  Unknown or Not Reported | 28 | 21 | 24 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 1 | 5
  Asian | 7 | 11 | 9 | 27
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Black or African American | 21 | 13 | 17 | 51
  White | 353 | 352 | 355 | 1060
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the number of months between study enrollment and death from any cause. Patients still alive at the last follow-up were censored on the date of last contact.
Time Frame: All patients were followed (with physical exams and histories) every three months for the first two years, then every six months for the next three years and then annually for the next five years.
Population: All randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel Poliglumex) | Arm II (Paclitaxel) | Arm III (Observation)
Number analyzed (Participants) | 387 | 384 | 386
Months | 60.0 [51.7 to 68.6] | 56.8 [47.3 to 65.9] | 58.3 [51.9 to 72.5]

2. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) was defined as the number of months between study enrollment and the date of first clinical, biochemical, or radiological evidence of progression or death due to any cause. Patients who were alive without progression at the time of analysis were censored on the date of the last tumor assessment.
Time Frame: Progression was assessed every 8 weeks for the first 15 months, then every 3 months, up to 14.2 years.
Population: All randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel Poliglumex) | Arm II (Paclitaxel) | Arm III (Observation)
Number analyzed (Participants) | 387 | 384 | 386
Months | 16.3 [14.4 to 18.9] | 18.9 [17.0 to 21.8] | 13.4 [11.2 to 15.7]

3. Secondary Outcome: Frequency and Severity of Adverse Effects Assessed by CTCAE v3.0
Description: Number of treated patients with Adverse Events (grade 3 or higher) observed while receiving randomized therapy among adverse event terms with at least 4 patients reporting.
Time Frame: Measured within 6 months of enrollment; through all cycles of chemotherapy and up to 30 days after the last cycle of chemotherapy. Up to 10 cycles of chemotherapy were allowed. Cycles were to be repeated every 3 weeks.
Population: Treated with randomized therapy
Measure: Number; unit: participants
Arm/Group | Arm I (Paclitaxel Poliglumex) | Arm II (Paclitaxel) | Arm III (Observation)
Number analyzed (Participants) | 379 | 374 | 386
participants
  Allergic Reaction / Hypersensitivity | 4 | 0 | 0
  Dehydration | 4 | 1 | 1
  Diarrhea | 7 | 3 | 2
  Dyspnea | 2 | 4 | 2
  Fatigue | 6 | 13 | 1
  Hemoglobin | 8 | 2 | 0
  Hyperglycemia | 5 | 6 | 1
  Hypertension | 2 | 4 | 5
  Hypokalemia | 9 | 2 | 0
  Leukocytes | 36 | 17 | 1
  Nausea | 7 | 3 | 4
  Neuropathy-Motor | 3 | 8 | 1
  Neutrophils | 82 | 62 | 2
  Obstruction, GI - Small Bowel Nos | 5 | 6 | 9
  Pain: Abdominal Pain Nos | 12 | 5 | 5
  Pain: Back | 7 | 4 | 1
  Pain: Extremity-Limb | 1 | 7 | 0
  Pain: Head/Headache | 4 | 2 | 0
  Pain: Joint | 5 | 3 | 1
  Thrombosis / Thrombus / Embolism | 5 | 4 | 2
  Vomiting | 8 | 6 | 3

4. Secondary Outcome: Patient-Reported Quality of Life (QOL)
Description: Patient reported quality of life was measured with the Treatment Outcome Index (TOI) of the Functional Assessment of Cancer Therapy for ovarian cancer (FACT-O TOI). The FACT-En TOI is a scale for assessing general QOL of ovarian cancer patients. The FACT-O TOI score ranges 0-100 with a large score suggesting better QOL.
Time Frame: 1. Prior to treatment 2. Prior to cycle 3 3. Prior to cycle 5 4. Prior to cycle 7 5. Prior to cycle 12 6. 12 months post treatment
Population: Provided baseline and >= 1 follow-up assessment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Paclitaxel Poliglumex) | Arm II (Paclitaxel) | Arm III (Observation)
Number analyzed (Participants) | 374 | 366 | 373
score on a scale
  Baseline | 78.2 (0.6) | 77.3 (0.7) | 77.4 (0.7)
  Prior to cycle 3 | 78.8 (0.7) | 76.9 (0.7) | 80.0 (0.7)
  Prior to cycle 5 | 79.3 (0.7) | 77.6 (0.7) | 80.8 (0.7)
  Prior to cycle 7 | 80.0 (0.7) | 77.5 (0.8) | 79.5 (0.8)
  Prior to cycle 12 | 78.3 (0.8) | 76.8 (0.8) | 79.2 (0.8)
  12 months post treatment | 78.8 (0.9) | 76.0 (0.9) | 77.4 (0.9)

5. Secondary Outcome: Patient-Reported Peripheral Neuropathy Symptoms
Description: Patient reported peripheral neuropathy symptoms was measured with the Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group - neurotoxicity subscale (short version) (FACT/GOG-Ntx subscale). The Ntx score ranges 0-16 with a large score suggesting less peripheral neuropathy symptoms.
Time Frame: as for outcome 4
Population: Provided baseline and >= 1 follow-up assessment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Paclitaxel Poliglumex) | Arm II (Paclitaxel) | Arm III (Observation)
Number analyzed (Participants) | 374 | 366 | 373
score on a scale
  Baseline | 11.4 (0.2) | 11.7 (0.2) | 11.8 (0.2)
  Prior to cycle 3 | 9.6 (0.2) | 10.6 (0.2) | 11.5 (0.2)
  Prior to cycle 5 | 9.5 (0.2) | 11.3 (0.2) | 11.9 (0.2)
  Prior to cycle 7 | 9.8 (0.2) | 11.3 (0.2) | 12.4 (0.2)
  Prior to cycle 12 | 9.4 (0.2) | 11.6 (0.2) | 12.2 (0.2)
  12 months post treatment | 10.7 (0.3) | 11.7 (0.3) | 12.4 (0.2)

ADVERSE EVENTS:
Time Frame: All patients were followed (with physical exams and histories) every three months for the first two years, then every six months for the next three years and then annually for the next 5 years.
Description: Eligible and treated participants were affected if they experienced grade 1-5 adverse event. As a point of clarification, for the all-cause mortality reporting, all of the enrolled patients were considered to be at risk. For the adverse event and serious adverse event reporting, only treated patients were considered to be at risk (i.e. ARM 1 (n=379), ARM 2 (n=374) ARM 3 (n=386)).
Arm/Group | Arm I (Paclitaxel Poliglumex) | Arm II (Paclitaxel) | Arm III (Observation)
All-Cause Mortality (participants affected / at risk) | 235/387 | 242/384 | 230/386
Serious Adverse Events (participants affected / at risk) | 50/379 | 39/374 | 1/386
Other Adverse Events (participants affected / at risk) | 378/379 | 372/374 | 312/386
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel Poliglumex) (N=379) | Arm II (Paclitaxel) (N=374) | Arm III (Observation) (N=386)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Rhinitis (Immune system disorders) | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Neutrophils (Blood and lymphatic system disorders) | 2 | 3 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0 | 0
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac General - Other (Cardiac disorders) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Weight Gain (General disorders) | 1 | 0 | 0
Fever (General disorders) | 2 | 0 | 0
Insomnia (General disorders) | 1 | 0 | 0
Nail Changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Obstruction, Gi - Stomach (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 0 | 3 | 0
Obstruction, Gi - Colon (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 2 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 4 | 6 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Dehydration (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 0 | 1 | 0
Febrile Neutropenia (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 1 | 0
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Pelvis Nos (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Wound (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Mood Alteration - Depression (Nervous system disorders) | 1 | 1 | 0
Mood Alteration - Anxiety (Nervous system disorders) | 1 | 1 | 0
Cns Ischemia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Neuropathy-Sensory (Nervous system disorders) | 0 | 1 | 0
Neuropathy-Motor (Nervous system disorders) | 1 | 2 | 0
Retinal Detachment (Eye disorders) | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0
Pain - Other (General disorders) | 1 | 0 | 0
Pain: Chest Wall (General disorders) | 0 | 0 | 1
Pain: Head/Headache (General disorders) | 2 | 0 | 0
Pain: Back (General disorders) | 1 | 0 | 0
Pain: Bone (General disorders) | 0 | 1 | 0
Pain: Stomach (General disorders) | 1 | 0 | 0
Pain: Abdominal Pain Nos (General disorders) | 1 | 0 | 0
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
2nd Mal: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Syndromes - Other (General disorders) | 0 | 1 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 4 | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel Poliglumex) (N=379) | Arm II (Paclitaxel) (N=374) | Arm III (Observation) (N=386)
Allergy/Immunology - Other (Immune system disorders) | 1 | 1 | 2
Allergic Reaction/Hypersensitivity (Immune system disorders) | 26 | 12 | 4
Rhinitis (Immune system disorders) | 19 | 31 | 19
Autoimmune Reaction (Immune system disorders) | 0 | 0 | 1
Otitis Middle Ear (Ear and labyrinth disorders) | 1 | 2 | 0
Auditory/Ear - Other (Ear and labyrinth disorders) | 1 | 3 | 2
Otitis External Ear (Ear and labyrinth disorders) | 1 | 0 | 1
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 5 | 4 | 5
Tinnitus (Ear and labyrinth disorders) | 23 | 29 | 14
Hearing (Monitoring Program) (Ear and labyrinth disorders) | 0 | 2 | 0
Neutrophils (Blood and lymphatic system disorders) | 190 | 213 | 28
Platelets (Blood and lymphatic system disorders) | 115 | 65 | 14
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 5 | 3 | 2
Bone Marrow Cellularity (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytes (Blood and lymphatic system disorders) | 229 | 231 | 44
Lymphopenia (Blood and lymphatic system disorders) | 5 | 10 | 2
Hemoglobin (Blood and lymphatic system disorders) | 270 | 283 | 83
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 8 | 10 | 4
Cardiac Arrhythmia - Other (Cardiac disorders) | 0 | 0 | 2
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 1 | 3 | 0
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 2 | 2 | 1
Vasovagal Episode (Cardiac disorders) | 0 | 0 | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0
Hypertension (Cardiac disorders) | 28 | 28 | 23
Valvular Heart Disease (Cardiac disorders) | 0 | 0 | 1
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 1 | 0 | 0
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 0 | 1
Cardiac General - Other (Cardiac disorders) | 5 | 2 | 1
Hypotension (Cardiac disorders) | 4 | 4 | 1
Inr (Vascular disorders) | 6 | 4 | 2
Coagulopathy - Other (Vascular disorders) | 1 | 0 | 2
Ptt (Vascular disorders) | 7 | 5 | 4
Constitutional Symptoms - Other (General disorders) | 3 | 6 | 6
Sweating (General disorders) | 5 | 14 | 7
Weight Gain (General disorders) | 45 | 46 | 27
Fever (General disorders) | 27 | 25 | 8
Weight Loss (General disorders) | 6 | 7 | 10
Hypothermia (General disorders) | 1 | 0 | 0
Rigors/Chills (General disorders) | 9 | 12 | 1
Fatigue (General disorders) | 254 | 277 | 143
Insomnia (General disorders) | 69 | 81 | 50
Nail Changes (Skin and subcutaneous tissue disorders) | 12 | 19 | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 135 | 239 | 76
Induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 4 | 6 | 6
Bruising (Skin and subcutaneous tissue disorders) | 13 | 13 | 10
Acne (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 50 | 46 | 20
Striae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 9 | 11 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 21 | 12
Burn (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 2 | 2
Flushing (Skin and subcutaneous tissue disorders) | 22 | 20 | 2
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 9 | 12 | 7
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Hot Flashes (Endocrine disorders) | 53 | 52 | 43
Diabetes (Endocrine disorders) | 3 | 1 | 3
Adh Secrection Abnormality (Endocrine disorders) | 0 | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Endocrine - Other (Endocrine disorders) | 2 | 2 | 1
Hypothyroidism (Endocrine disorders) | 3 | 1 | 3
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 7 | 11 | 13
Ulcer,gi - Esophagus (Gastrointestinal disorders) | 1 | 0 | 0
Dental: Periodontal (Gastrointestinal disorders) | 2 | 1 | 0
Obstruction, Gi - Colon (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 5 | 3
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 5 | 4 | 3
Heartburn (Gastrointestinal disorders) | 35 | 32 | 19
Dental: Teeth (Gastrointestinal disorders) | 2 | 7 | 0
Mucositis (Functional/Sympt) - Pharynx (Gastrointestinal disorders) | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 2 | 0
Dental: Teeth Development (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 5 | 4 | 1
Distention (Gastrointestinal disorders) | 25 | 23 | 34
Taste Alteration (Gastrointestinal disorders) | 11 | 19 | 2
Incontinence, Anal (Gastrointestinal disorders) | 2 | 5 | 2
Dry Mouth (Gastrointestinal disorders) | 3 | 7 | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 6 | 15 | 2
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 3 | 1 | 11
Obstruction, Gi - Jejunum (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 15 | 21 | 1
Vomiting (Gastrointestinal disorders) | 53 | 41 | 36
Anorexia (Gastrointestinal disorders) | 41 | 46 | 21
Dehydration (Gastrointestinal disorders) | 5 | 3 | 3
Constipation (Gastrointestinal disorders) | 156 | 158 | 88
Nausea (Gastrointestinal disorders) | 145 | 137 | 63
Gastrointestinal - Other (Gastrointestinal disorders) | 9 | 10 | 9
Diarrhea (Gastrointestinal disorders) | 88 | 97 | 56
Prolapse Of Stoma, Gi (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage, Gu - Stoma (Vascular disorders) | 1 | 0 | 0
Hemorrhage, Gu - Vagina (Vascular disorders) | 9 | 6 | 1
Hemorrhage, Gu - Urethra (Vascular disorders) | 0 | 1 | 0
Hemorrhage, Gi - Rectum (Vascular disorders) | 6 | 5 | 5
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 0 | 1 | 0
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 19 | 8 | 1
Hematoma (Vascular disorders) | 3 | 1 | 0
Hemorrhage, Gi - Anus (Vascular disorders) | 1 | 1 | 0
Hemorrhage, Gi - Esophagus (Vascular disorders) | 0 | 0 | 1
Hemorrhage, Gi - Lower Gi Nos (Vascular disorders) | 0 | 1 | 0
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 3 | 1 | 0
Hemorrhage, Gu - Bladder (Vascular disorders) | 0 | 3 | 2
Petechiae (Vascular disorders) | 1 | 0 | 0
Hemorrhage/Bleeding - Other (Vascular disorders) | 3 | 1 | 1
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 1 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Liver Dysfunction (Hepatobiliary disorders) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 13 | 12 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Nose (Infections and infestations) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Lip/Perioral (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 3 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Eye Nos (Infections and infestations) | 0 | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Soft Tissue Nos (Infections and infestations) | 3 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Peristomal (Infections and infestations) | 1 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 2 | 1 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 2 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Otitis Media Nos (Infections and infestations) | 2 | 5 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 3 | 5 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lip/Perioral (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Nerve-Peripheral (Infections and infestations) | 0 | 0 | 1
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 3 | 1
Inf Unknown Anc: Sinus (Infections and infestations) | 4 | 6 | 6
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 2 | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Colon (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 13 | 16 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 3 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Ungual (Nails) (Infections and infestations) | 1 | 0 | 1
Inf Unknown Anc: Stomach (Infections and infestations) | 0 | 1 | 0
Infection - Other (Infections and infestations) | 9 | 16 | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Nerve-Peripheral (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Vulva (Infections and infestations) | 0 | 0 | 1
Inf Unknown Anc: Vagina (Infections and infestations) | 1 | 2 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 5 | 1 | 1
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 2 | 1 | 3
Inf Unknown Anc: Upper Aerodigestive (Infections and infestations) | 0 | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Pharynx (Infections and infestations) | 0 | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 3 | 4 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 6 | 5 | 5
Inf Unknown Anc: Pharynx (Infections and infestations) | 0 | 0 | 1
Inf Unknown Anc: Bronchus (Infections and infestations) | 1 | 0 | 1
Inf Unknown Anc: Eye Nos (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Joint (Infections and infestations) | 0 | 0 | 1
Inf Unknown Anc: Lymphatic (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 7 | 8 | 3
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 4 | 4 | 3
Inf Unknown Anc: Wound (Infections and infestations) | 0 | 0 | 2
Inf Unknown Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Foreign Body (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Dental-Tooth (Infections and infestations) | 0 | 0 | 1
Inf Unknown Anc: Appendix (Infections and infestations) | 0 | 0 | 1
Inf Unknown Anc: Anal/Perianal (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Abdomen Nos (Infections and infestations) | 1 | 1 | 0
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1 | 1 | 4
Inf Unknown Anc: Peristomal (Infections and infestations) | 0 | 0 | 1
Inf Unknown Anc: Middle Ear (Infections and infestations) | 0 | 1 | 1
Inf Unknown Anc: External Ear (Infections and infestations) | 1 | 2 | 1
Inf W/Gr 3 Or 4 Anc: Pelvis Nos (Infections and infestations) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Upper Airway Nos (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Sinus (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 3 | 6 | 3
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 1 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Catheter-Related (Infections and infestations) | 1 | 0 | 0
Lymphatics - Other (Blood and lymphatic system disorders) | 3 | 2 | 0
Lymphocele (Blood and lymphatic system disorders) | 0 | 0 | 1
Edema: Viscera (Blood and lymphatic system disorders) | 0 | 1 | 0
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 2 | 5 | 2
Edema: Limb (Blood and lymphatic system disorders) | 72 | 70 | 31
Edema: Head And Neck (Blood and lymphatic system disorders) | 5 | 7 | 5
Dermal Change (Blood and lymphatic system disorders) | 0 | 0 | 1
Ast (Metabolism and nutrition disorders) | 69 | 24 | 12
Gfr (Metabolism and nutrition disorders) | 2 | 4 | 3
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 12 | 13 | 4
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Cholesterol,serum High (Metabolism and nutrition disorders) | 6 | 6 | 4
Proteinuria (Metabolism and nutrition disorders) | 1 | 0 | 0
Hemoglobinuria (Metabolism and nutrition disorders) | 0 | 0 | 1
Creatinine (Metabolism and nutrition disorders) | 14 | 21 | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 | 12 | 6
Alt (Metabolism and nutrition disorders) | 36 | 27 | 8
Alkaline Phosphatase (Metabolism and nutrition disorders) | 38 | 32 | 16
Bilirubin (Metabolism and nutrition disorders) | 6 | 2 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 4 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 22 | 15 | 8
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 0 | 1 | 1
Amylase (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 5 | 9 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 15 | 10 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 6 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 79 | 67 | 27
Hypokalemia (Metabolism and nutrition disorders) | 33 | 28 | 13
Hypoglycemia (Metabolism and nutrition disorders) | 10 | 14 | 9
Hypercalcemia (Metabolism and nutrition disorders) | 13 | 11 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 37 | 29 | 10
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 10 | 12 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Joint-Function (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7
Gait/Walking (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 15 | 13 | 14
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 10 | 16 | 11
Muscle Weakness - Trunk (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle Weakness - Left-Sided (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle Weakness - Facial (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 6 | 10 | 9
Syncope (Nervous system disorders) | 2 | 1 | 1
Involuntary Movement (Nervous system disorders) | 1 | 4 | 1
Psychosis (Nervous system disorders) | 0 | 1 | 0
Neurology - Other (Nervous system disorders) | 1 | 8 | 5
Mental Status (Nervous system disorders) | 1 | 0 | 1
Mood Alteration - Depression (Nervous system disorders) | 44 | 62 | 47
Mood Alteration - Anxiety (Nervous system disorders) | 43 | 53 | 43
Mood Alteration - Agitation (Nervous system disorders) | 6 | 10 | 1
Tremor (Nervous system disorders) | 3 | 2 | 2
Speech Impairment (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1
Personality (Nervous system disorders) | 2 | 0 | 0
Irritability (Nervous system disorders) | 0 | 3 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1
Cognitive Disturbance (Nervous system disorders) | 7 | 5 | 1
Ataxia (Nervous system disorders) | 4 | 5 | 1
Confusion (Nervous system disorders) | 2 | 3 | 0
Memory Impairment (Nervous system disorders) | 17 | 37 | 14
Dizziness (Nervous system disorders) | 38 | 42 | 17
Neuropathy,cranial - Cn Viii Hearing/Balance (Nervous system disorders) | 1 | 0 | 0
Neuropathy,cranial - Cn V Motor-Jaw Muscles (Nervous system disorders) | 0 | 1 | 1
Neuropathy-Sensory (Nervous system disorders) | 318 | 294 | 175
Neuropathy-Motor (Nervous system disorders) | 33 | 31 | 15
Ocular/Visual - Other (Eye disorders) | 4 | 9 | 1
Nystagmus (Eye disorders) | 0 | 0 | 1
Watery Eye (Eye disorders) | 0 | 5 | 0
Glaucoma (Eye disorders) | 1 | 1 | 0
Dry Eye (Eye disorders) | 2 | 5 | 2
Ocular Surface Disease (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 2 | 2 | 1
Photophobia (Eye disorders) | 1 | 1 | 2
Flashing Lights/Floaters (Eye disorders) | 3 | 5 | 3
Diplopia (Eye disorders) | 0 | 1 | 0
Blurred Vision (Eye disorders) | 19 | 30 | 12
Eyelid Dysfunction (Eye disorders) | 0 | 1 | 1
Pain - Other (General disorders) | 19 | 24 | 22
Pain: Urethra (General disorders) | 9 | 2 | 2
Pain: Perineum (General disorders) | 0 | 2 | 0
Pain: Pelvis (General disorders) | 20 | 14 | 18
Pain: Breast (General disorders) | 7 | 2 | 3
Pain: Vagina (General disorders) | 3 | 7 | 7
Pain: Chest /Thorax Nos (General disorders) | 21 | 18 | 7
Pain: Chest Wall (General disorders) | 12 | 4 | 3
Pain: Throat/Pharynx/Larynx (General disorders) | 6 | 18 | 0
Pain: Pleura (General disorders) | 3 | 0 | 1
Pain: Eye (General disorders) | 1 | 3 | 0
Pain: Head/Headache (General disorders) | 62 | 52 | 22
Pain: Neck (General disorders) | 6 | 7 | 7
Pain: Intestine (General disorders) | 2 | 1 | 0
Pain: Extremity-Limb (General disorders) | 61 | 76 | 30
Pain: Buttock (General disorders) | 1 | 2 | 0
Pain: Back (General disorders) | 52 | 52 | 48
Pain: Joint (General disorders) | 106 | 133 | 81
Pain: Bone (General disorders) | 21 | 25 | 9
Pain: Gallbladder (General disorders) | 1 | 0 | 1
Pain: Kidney (General disorders) | 0 | 2 | 0
Pain: Bladder (General disorders) | 1 | 6 | 2
Pain: Pain Nos (General disorders) | 5 | 7 | 2
Pain: Stomach (General disorders) | 6 | 5 | 1
Pain: Rectum (General disorders) | 0 | 1 | 2
Pain: Oral Cavity (General disorders) | 1 | 1 | 1
Pain: Dental/Teeth/Peridontal (General disorders) | 4 | 6 | 2
Pain: Abdominal Pain Nos (General disorders) | 111 | 102 | 120
Pain: Scalp (General disorders) | 0 | 1 | 0
Pain: Oral - Gums (General disorders) | 0 | 2 | 0
Pain: Skin (General disorders) | 0 | 1 | 0
Pain: Lip (General disorders) | 1 | 1 | 0
Pain: Middle Ear (General disorders) | 2 | 3 | 3
Pain: External Ear (General disorders) | 1 | 3 | 0
Pain: Cardiac/ Heart (General disorders) | 2 | 0 | 1
Pain: Face (General disorders) | 1 | 2 | 0
Pain: Liver (General disorders) | 1 | 0 | 0
Pain: Muscle (General disorders) | 77 | 102 | 44
Pain: Anus (General disorders) | 1 | 0 | 1
Pain: Neuralgia (General disorders) | 7 | 9 | 1
Pain: Sinus (General disorders) | 1 | 3 | 0
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 2
Airway Obstruction - Bronchus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 11 | 13 | 6
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 75 | 31
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 66 | 72 | 41
Renal/Genitourinary - Other (Renal and urinary disorders) | 7 | 4 | 3
Leak, Gu - Bladder (Renal and urinary disorders) | 3 | 0 | 0
Cystitis (Renal and urinary disorders) | 3 | 2 | 4
Urinary Color Change (Renal and urinary disorders) | 0 | 3 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 2 | 3
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1 | 0 | 1
Incontinence, Urinary (Renal and urinary disorders) | 16 | 19 | 13
Bladder Spasm (Renal and urinary disorders) | 1 | 4 | 3
Urinary Frequency (Renal and urinary disorders) | 15 | 30 | 24
2nd Mal: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Libido (Reproductive system and breast disorders) | 5 | 2 | 6
Vaginal Dryness (Reproductive system and breast disorders) | 11 | 9 | 8
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 2 | 1 | 3
Vaginitis (Reproductive system and breast disorders) | 3 | 6 | 5
Vaginal Stenosis (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 4 | 9 | 4
Intra-Op Injury: Abdomen Nos (Surgical and medical procedures) | 1 | 0 | 0
Flu-Like Syndrome (General disorders) | 6 | 6 | 3
Vascular - Other (Vascular disorders) | 1 | 2 | 1
Vein Injury - Extremity-Lower (Vascular disorders) | 0 | 1 | 0
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 0 | 2 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2 | 3 | 2
Phlebitis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT00108745/Prot_SAP_000.pdf